CLINICAL TRIAL: NCT01464710
Title: Genetic Assessment of Early to Late macuLar dEgeneration studY 2
Brief Title: Genetic Assessment of Early to Late Macular Degeneration Study
Acronym: GALLEY2
Status: Completed | Type: Observational
Sponsor: Henry Ferreyra (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Henry Ferreyra, Principal Investigator, University of California, San Diego
Organization: University of California, San Diego (Other)
Other Study IDs: 080585
Record Dates: First submitted 2011-10-31; First posted 2011-11-03 (Estimated); Last update posted 2019-06-21 (Actual); Status verified 2019-06

CONDITIONS: Age-related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Specimen collected for genotype analysis.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to determine if polymorphisms at rs11200638 on HTRA1 and rs1061170 on CFH are associated with an accelerated progression to advanced AMD (wet AMD or GA) in patients with early AMD (soft confluent drusen>120 microns ) in the study eye, and with either early AMD or advanced AMD in the non-study eye.

DETAILED DESCRIPTION:
Age-related macular degeneration (AMD) is the leading cause of blindness in the developed world. To date, two major polymorphisms on the HTRA1 and CFH genes have been associated with AMD. Progression and vision loss need to be followed and treated promptly in order to preserve vision. This study will provide more information on the genetics of disease progression and may lead to future guidelines for patient follow-up and treatment.

This study consists of a blood draw and observation of eye conditions. Consented, enrolled patients will come in every four months as per standard of care. At each visit, visual acuity measurement, slit lamp exam, indirect ophthalmoscopy, fundus photos, and spectral domain optical coherence tomography will be performed. Every 8 months, or per standard of care, fluoroscein angiography will be performed. DNA extraction and genotyping will be performed, and correlations between HTRA1 and CFH genotypes and the progression to bilateral advanced AMD will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be eligible if the following criteria are met:
* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age > 45 years
* Disease related considerations
* Subjects with a diagnosis of advanced AMD in one eye (either CNV or geographic atrophy) and soft confluent drusen in the study eye OR subjects with bilateral large soft drusen.

Exclusion Criteria:

* Subjects with any other progressive retinal disease that may impair the physician's ability to assess the severity of AMD

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with a diagnosis of advanced AMD in one eye (either CNV or geographic atrophy) and soft confluent drusen in the study eye OR subjects with bilateral large soft drusen.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2008-04; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
To determine the allele frequency for patients that progress to bilateral advanced AMD in the study eye | 5 years

SECONDARY OUTCOMES:
To determine the allele frequency for patients that do not progress to bilateral advanced AMD in the study eye. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Henry Ferreyra, M.D, Study Chair — University of California, San Diego
Locations (3):
- United States (3):
  - University of California, San Diego, La Jolla, California
  - California Retina Consultants, Santa Barbara, California
  - Medical Center Ophthalmology Associates, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No
Data not available.